CLINICAL TRIAL: NCT02444897
Title: The Comparison Between Epidural and Intravenous Patient-controlled Analgesia for Laparoscopic Gastrectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Seung Wan Ryu, Director of Gastrointesinal surgery, associate professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012-12-514
Record Dates: First submitted 2015-04-25; First posted 2015-05-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; epidural; PCA; laparoscopy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidural PCA group (Experimental): Epidural patient-controlled analgesia group
  Interventions: Drug: Epidural PCA Ropivacaine
- IV PCA group (Active Comparator): Intravenous patient-controlled analgesia
  Interventions: Drug: IV PCA Fentanyl+nefopam+Ramosetron

INTERVENTIONS:
Drug: Epidural PCA Ropivacaine — Epidural catheter insertion at T10 level before surgery, the tip of catheter location at T8-9 level.
  Total volume: 500ml, 16.7mcg/kg+0.75% Ropivacaine 80ml+N/S
  Other Names: Epidural patient-controlled analgesia Ropivacaine
  Arms: Epidural PCA group
Drug: IV PCA Fentanyl+nefopam+Ramosetron — Total volume: 84ml, Fentanyl 1000mcg+nefopam 120mg+Ramosetron 0.3mg Basal infusion: 1ml/hr, Bolus: 0.5ml with a lockout time 15min.
  Other Names: intravenous patient-controlled analgesia
  Arms: IV PCA group

SUMMARY:
This study was designed to assess the effectiveness of epidural patient-controlled analgesia compared to intravenous patient-controlled analgesia in patients undergoing laparoscopic gastrectomy. The investigators hypothesized that epidural PCA would be more effective in pain control than IV PCA even for laparoscopic gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma in stomach
* Males or Females, aged≥19 years and ≤80 years
* Scheduled as laparoscopic gastrectomy
* Patient has given their written informed consent to participate in the study

Exclusion Criteria:

* History of hypersensitivity for analgesics
* Recent history of narcotic analgesics
* Disability of central nerve system
* Uncontrolled co-morbidity

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
VAS score | 24 hours after operation
  pain degree was checked at every 24hours for 5days after operation

SECONDARY OUTCOMES:
number of participants with complication | for 5days after operation
  PCA related complication
Bowel motility | for 5days after operation
  by counting Colomark on abdomen x-ray

CONTACTS AND LOCATIONS:
Overall Officials: Seung Wan Ryu, M.D., Ph.D., Principal Investigator — Director of gastrointestinal surgery devision, associate proffessor
Locations (1):
- Keimyung University Dongsan Medical Center, Daegu, South Korea